CLINICAL TRIAL: NCT00383240
Title: A 26-Week Placebo-Controlled Efficacy and Safety Study of Mometasone Furoate/Formoterol Fumarate Combination Formulation Compared With Mometasone Furoate and Formoterol Monotherapy in Subjects With Persistent Asthma Previously Treated With Medium-Dose Inhaled Glucocorticosteroids
Brief Title: Effects of Mometasone Furoate/Formoterol Combination Versus Mometasone Furoate Alone in Persistent Asthmatics (Study P04334AM1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04334; EUDRACT No.: 2006-001578-25;
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; BID protein, human; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MF/F MDI 200/10 mcg BID (Experimental)
  Interventions: Drug: mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID
- MF MDI 200 mcg BID (Experimental)
  Interventions: Drug: Mometasone furoate MDI (MF MDI) 200 mcg
- F MDI 10 mcg BID (Experimental)
  Interventions: Drug: formoterol fumarate 10 mcg
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID — MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 26 weeks
  Other Names: SCH 418131
  Arms: MF/F MDI 200/10 mcg BID
Drug: Mometasone furoate MDI (MF MDI) 200 mcg — MF 200 mcg via metered dose inhaler twice daily for 26 weeks
  Other Names: SCH 32088
  Arms: MF MDI 200 mcg BID
Drug: formoterol fumarate 10 mcg — F via metered dose inhaler 10 mcg twice a day for 26 weeks
  Other Names: Foradil
  Arms: F MDI 10 mcg BID
Drug: Placebo — Placebo metered dose inhaler twice a day for 26 weeks
  Arms: Placebo BID

SUMMARY:
This is a randomized, multi-center, double-blind, double-dummy, placebo-controlled, parallel-group study, evaluating the efficacy of mometasone furoate (MF) /formoterol fumarate (F)[MF/F] metered dose inhaler (MDI) versus MF for 26 weeks. Prior to the 26-week double-blind Treatment Period, subjects will receive open-label MF MDI 200 mcg twice daily (BID) for 2 to 3 weeks during the Run-in Period. Efficacy will be measured by The Area Under the Curve From 0 to 12 Hours [AUC](0-12 hours) of the Change From Baseline to the Week 12 Endpoint

in Forced Expiratory Volume in One Second (FEV1) [Time Frame: Baseline to Week 12] and Time-to-First Severe Asthma Exacerbation across the 26-week treatment period.

ELIGIBILITY:
Adult and adolescent subjects of either sex and any race, at least 12 years of age or older, with a diagnosis of asthma of at least 12 months' duration, will be eligible for enrollment. Subjects must meet all of the inclusion criteria and none of the exclusion criteria to receive treatment assignment.

Key Inclusion Criteria Include

- A subject must have been using a medium daily dose of inhaled glucocorticosteroid (ICS) (either alone or in combination with a long-acting beta agonist (LABA)) for at least 12 weeks and must have been on a stable regimen (daily dose unchanged) for at least 2 weeks prior to Screening. Medium daily doses of ICS are defined as follows:

* >500 to 1000 mcg beclomethasone chlorofluorocarbon (CFC)
* >250 to 500 mcg beclomethasone hydrofluoroalkane (HFA)
* >600 to 1000 mcg budesonide dry powder inhaler (DPI)
* >1000 to 2000 mcg flunisolide
* >250 to 500 mcg fluticasone
* 400 mcg MF
* >1000 to 2000 mcg triamcinolone acetonide

Note: Dose delivery by method or modality other than those noted above must be equivalent.

* If, based upon the medical judgment of the investigator, there is no inherent harm in changing the subject's current asthma therapy, then the subject (and parent/guardian, if applicable) must be willing to discontinue his/her prescribed ICS or ICS/LABA combination at the Screening Visit, and be transferred to open-label treatment with MF MDI 200 mcg BID for 2 to 3 weeks prior to the Baseline/Randomization Visit.
* To document the diagnosis of asthma and assure the subject's responsiveness to bronchodilators before randomization one of the following methods can be used at the Screening Visit, Day -14, or thereafter, but prior to the Baseline Visit:

  1. The subject must demonstrate an increase in absolute FEV1 of at least 12% and at least 200 mL within 15 minutes after administration of four inhalations of albuterol/salbutamol (total dose of 360 to 400 mcg) or of nebulized SABA (2.5 mg) if confirmed as standard office practice, OR
  2. The subject must demonstrate a peak expiratory flow (PEF) variability of more than 20% expressed as a percentage of the highest and lowest morning prebronchodilator PEF over at least 1 week, OR
  3. The subject must demonstrate a diurnal variation in PEF of more than 20% based on the difference between the prebronchodilator morning value and the postbronchodilator value from the evening before, expressed as a percentage of the mean daily PEF value.
* At the Screening Visit, the subject's FEV1 must be ≥60% and ≤90% predicted.
* At the Baseline Visit, the subject's FEV1 must be ≥60% and ≤85% predicted when all restricted medications have been withheld for the appropriate intervals.
* Clinical laboratory tests (complete blood counts [CBC], blood chemistries, and urinalysis) conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor. An electrocardiogram (ECG) using a centralized trans-telephonic technology at the Screening Visit must be clinically acceptable to the investigator. A chest x-ray performed at the Screening Visit, or within 12 months prior to the Screening Visit, must be clinically acceptable to the investigator.
* A female subject of childbearing potential must have been using a medically acceptable, adequate form of birth control. This includes: 1) hormonal contraceptives as prescribed by a physician (oral combined, hormonal implant); 2) medically prescribed intra-uterine device (IUD); 3) condom in combination with a spermicide (double barrier method); 4) monogamous relationship with a male partner who has had a vasectomy. The subject must have started this birth control method at least 3 months prior to Screening (with the exception of condom in combination with spermicide), and must agree to continue its use for the duration of the study. A female subject of childbearing potential who is not currently sexually active must agree and consent to using a medically acceptable birth control method should she become sexually active during the course of this study. Women who have been surgically sterilized or are at least 1 year postmenopausal are not considered to be of childbearing potential. A female subject of childbearing potential must have a negative serum pregnancy test at Screening in order to be considered eligible for enrollment.

Key Exclusion Criteria Include

* A subject who demonstrates a change (increase or decrease) in absolute FEV1 of >20% at any time from the Screening Visit up to and including the Baseline Visit.
* A subject who requires the use of greater than eight inhalations per day of SABA MDI, or two or more nebulized treatments per day of 2.5 mg SABA, on any 2 consecutive days from the Screening Visit up to and including the Baseline Visit.
* A subject who experiences a decrease in AM or PM PEF below the Screening Period stability limit on any 2 consecutive days prior to Randomization.
* A subject who experiences an occurrence of any clinical deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication (other than SABA) as judged by the clinical investigator at any time from the Screening Visit up to and including the Baseline Visit.
* A subject who is a smoker or ex-smoker and has smoked within the previous year or has had a cumulative smoking history >10 pack-years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nathan RA, Nolte H, Pearlman DS; P04334 Study Investigators. Twenty-six-week efficacy and safety study of mometasone furoate/formoterol 200/10 microg combination treatment in patients with persistent asthma previously receiving medium-dose inhaled corticosteroids. Allergy Asthma Proc. 2010 Jul-Aug;31(4):269-79. doi: 10.2500/aap.2010.31.3364. Epub 2010 Jul 30. PMID 20678306

RESULTS

PARTICIPANT FLOW:
Groups:
- MF/F MDI 200/10 mcg BID: mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) 200/10 mcg twice daily (BID) for 26 weeks
- MF MDI 200 mcg BID: Mometasone furoate (MF) MDI 200 mcg BID for 26 weeks
- F MDI 10 mcg BID: Formoterol fumarate (F) MDI 10 mcg BID for 26 weeks
- Placebo BID: Placebo MDI BID for 26 weeks
Period: Overall Study
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Started | 191 | 192 | 202 | 196
Completed | 156 | 159 | 117 | 119
Not Completed | 35 | 33 | 85 | 77
Not completed — Adverse Event | 4 | 6 | 9 | 7
Not completed — Treatment Failure | 8 | 13 | 47 | 46
Not completed — Lost to Follow-up | 3 | 0 | 0 | 2
Not completed — Withdrawal by subject, reasons unrelated | 6 | 3 | 8 | 8
Not completed — Withdrawal by subjects, reasons related | 0 | 1 | 3 | 5
Not completed — Protocol Violation | 4 | 5 | 9 | 6
Not completed — Did not meet protocol eligibility | 9 | 4 | 9 | 3
Not completed — Administrative | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID | Total
Number analyzed (Participants) | 191 | 192 | 202 | 196 | 781
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 10 | 18 | 16 | 63
  Between 18 and 65 years | 161 | 173 | 174 | 169 | 677
  >=65 years | 11 | 9 | 10 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (16.3) | 42.8 (14.9) | 41.9 (15.3) | 41.9 (15.3) | 42.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 112 | 129 | 122 | 460
  Male | 94 | 80 | 73 | 74 | 321

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Time Curve From 0 to 12 Hours (AUC(0-12 Hours)) of Change From Baseline to Week 12 in Forced Expiratory Volume (Liters) in 1 Second (FEV1) for MF/F Versus MF
Time Frame: Baseline to Endpoint (12 weeks)
Population: Intent to Treat (ITT) population
Measure: Least Squares Mean (Standard Deviation); unit: liters x hours
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 190 | 190 | 202 | 193
liters x hours
  Baseline (n=188/189/198/192, respectively) | 3.20 (2.96) | 1.29 (2.96) | 2.73 (2.96) | 1.42 (2.96)
  Endpoint (Change from Baseline) | 3.19 (3.98) | 1.31 (3.98) | 1.60 (3.98) | 0.51 (3.98)
Statistical Analysis 1: Comparison: MF/F MDI 200/10 mcg BID vs MF MDI 200 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 3: Comparison: MF/F MDI 200/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 4: Comparison: MF MDI 200 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p = 0.491, ANCOVA — P-Value for Endpoint
Statistical Analysis 5: Comparison: MF MDI 200 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.055, ANCOVA — P-Value for Endpoint
Statistical Analysis 6: Comparison: F MDI 10 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.008, ANCOVA — P-Value for Endpoint

2. Secondary Outcome: Change From Baseline to Week 26 in Asthma Quality of Life Questionnaire With Standardized Activities (AQLQ[S]) Total Score
Description: AQLQ(S) consists of 32 questions each scaled from 1 (worst case) to 7 (best case). Standard deviations are pooled.
Time Frame: Baseline to Week 26
Population: ITT population with non-missing post-baseline AQLQ result
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 183 | 189 | 187 | 189
units on a scale
  Baseline (n=183/189/187/189, respectively) | 5.38 (1.10) | 5.40 (1.13) | 5.51 (1.11) | 5.56 (1.06)
  Change from Baseline to Endpoint (26 weeks) | 0.49 (0.85) | 0.37 (0.85) | 0.05 (0.85) | -0.01 (0.85)
Statistical Analysis 1: Comparison: MF/F MDI 200/10 mcg BID vs MF MDI 200 mcg BID; Test type: Superiority or Other; p = 0.174, ANCOVA — P-Value for Endpoint
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 3: Comparison: MF/F MDI 200/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 4: Comparison: MF MDI 200 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 5: Comparison: MF MDI 200 mcg BID vs Placebo BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 6: Comparison: F MDI 10 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.521, ANCOVA — P-Value for Endpoint

3. Primary Outcome: Time-to-first Asthma Exacerbation Over the 26-week Treatment Period for the Comparison of MF/F Versus F
Description: This endpoint was to measure the time it took for 50% of subjects in a treatment arm to experience a severe asthma exacerbation (also see the posted Other Pre-specified Outcome: Number of Participants With at Least One Severe Asthma Exacerbation)
Time Frame: 26-week Treatment Period
Population: All Randomized Subjects
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 191 | 192 | 202 | 196
days | NA (NA) [NA to NA] — Since less than 50% of the subjects in the MF/F and MF treatment groups experienced an asthma exacerbation by the end of the 26 week treatment period, median time-to-first asthma exacerbation can not be determined but is at least 26 weeks. | NA (NA) [NA to NA] — Since less than 50% of the subjects in the MF/F and MF treatment groups experienced an asthma exacerbation by the end of the 26 week treatment period, median time-to-first asthma exacerbation can not be determined but is at least 26 weeks. | 92 (NA) [24 to NA] — In the F treatment group a subject experienced an asthma exacerbation on day 193 since the event was observed on the final visit performed 10 days beyond the scheduled 26-week treatment period schedule. Therefore the InterQuartile Range is 24 to 193. | 131 (NA) [25 to NA] — Since less than 75% of the subjects in the placebo group experienced an asthma exacerbation by the end of the 26 week treatment period, 3rd quartile time-to-first asthma exacerbation can not be determined but is at least 26 weeks.

4. Secondary Outcome: Change From Baseline to Week 26 in the Asthma Control Questionnaire (ACQ) Score
Description: ACQ consists of seven questions each scaled from 0 (best case) to 6 (worst case).
Time Frame: Baseline to week 26
Population: ITT population with non-missing post-baseline ACQ result
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 179 | 186 | 184 | 187
units on a scale
  Baseline (n=179/186/184/187, respectively) | 1.47 (0.75) | 1.46 (0.77) | 1.43 (0.79) | 1.41 (0.75)
  Change from Baseline to Endpoint (week 26) | -0.40 (0.74) | -0.23 (0.74) | 0.11 (0.74) | 0.14 (0.74)
Statistical Analysis 1: Comparison: MF/F MDI 200/10 mcg BID vs MF MDI 200 mcg BID; Test type: Superiority or Other; p = 0.026, ANCOVA — P-Value for Endpoint
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 3: Comparison: MF/F MDI 200/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 4: Comparison: MF MDI 200 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 5: Comparison: MF MDI 200 mcg BID vs Placebo BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 6: Comparison: F MDI 10 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.738, ANCOVA — P-Value for Endpoint

5. Secondary Outcome: Change From Baseline in Proportion of Nights Across the Treatment Period With Nocturnal Awakenings Due to Asthma Which Require Use of Short-acting Beta 2-agonist (SABA)
Description: Baseline is the proportion of nights of last week (Days -7 to 1) prior to first dose with nocturnal awakenings. Scale is measured as 0 to 1 with 0=no awakenings to 1=awakenings every night. Standard deviation is pooled.
Time Frame: Baseline to Endpoint
Population: ITT population from the entire 26-week treatment period
Measure: Least Squares Mean (Standard Deviation); unit: Ratio
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 186 | 191 | 199 | 194
Ratio
  Baseline (n=186/191/199/194, respectively) | 0.18 (0.31) | 0.16 (0.27) | 0.16 (0.27) | 0.15 (0.27)
  Change from Baseline to Endpoint | -0.08 (0.17) | -0.05 (0.17) | 0.01 (0.17) | 0.00 (0.17)
Statistical Analysis 1: Comparison: MF/F MDI 200/10 mcg BID vs MF MDI 200 mcg BID; Test type: Superiority or Other; p = 0.063, ANCOVA — P-Value for endpoint
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 3: Comparison: MF/F MDI 200/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 4: Comparison: MF MDI 200 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p < .001, ANCOVA — P-Value for Endpoint
Statistical Analysis 5: Comparison: MF MDI 200 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.003, ANCOVA — P-Value for Endpoint
Statistical Analysis 6: Comparison: F MDI 10 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.601, ANCOVA — P-Value for Endpoint

6. Other Pre Specified Outcome: Number of Participants With at Least One Severe Asthma Exacerbation
Description: A severe asthma exacerbation was defined as a clinically judged deterioration of asthma or a meaningful reduction in lung function based on any of the following criteria during the Treatment Period:
  * A decrease in FEV1 below the Treatment Period stability limit at any visit,
  * A decrease in AM or PM peak flow below the Treatment Period stability limits on any 2 consecutive days,
  * An occurrence of any clinical deterioration of asthma (ie, asthma attack) that resulted in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication.
Time Frame: Baseline to Week 26
Population: All Randomized Subjects
Measure: Number; unit: participants
Arm/Group | MF/F MDI 200/10 mcg BID | MF MDI 200 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 191 | 192 | 202 | 196
participants | 58 | 65 | 109 | 109

ADVERSE EVENTS:
Groups:
- OL MF MDI 200 MCG BID: Participants received 2 to 3 weeks (approximately) of open-label (OL), run-in medication with MF MDI 200 mcg BID prior to the 26-week double-blind treatment period.
Arm/Group | OL MF MDI 200 MCG BID | MF/F MDI 200/10 MCG BID | MF MDI 200 MCG BID | F MDI 10 MCG BID | PLACEBO
Serious Adverse Events (participants affected / at risk) | 4/984 | 5/191 | 3/192 | 3/202 | 3/196
Other Adverse Events (participants affected / at risk) | 25/984 | 31/191 | 35/192 | 29/202 | 30/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL MF MDI 200 MCG BID (N=984) | MF/F MDI 200/10 MCG BID (N=191) | MF MDI 200 MCG BID (N=192) | F MDI 10 MCG BID (N=202) | PLACEBO (N=196)
DENGUE FEVER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL DECOMPRESSION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL MF MDI 200 MCG BID (N=984) | MF/F MDI 200/10 MCG BID (N=191) | MF MDI 200 MCG BID (N=192) | F MDI 10 MCG BID (N=202) | PLACEBO (N=196)
NASOPHARYNGITIS (Infections and infestations) | 8 (8) | 12 (13) | 15 (22) | 13 (14) | 7 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (7) | 11 (13) | 16 (16) | 12 (16) | 17 (17)
HEADACHE (Nervous system disorders) | 11 (13) | 9 (10) | 10 (17) | 6 (8) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less